CLINICAL TRIAL: NCT02580708
Title: A Phase 1/2 Study of the Safety and Efficacy of Rociletinib When Administered in Combination With Trametinib in Patients With Activating EGFR Mutation-positive Advanced or Metastatic Non-small Lung Cancer (NSCLC)
Brief Title: Phase 1/2 Study of the Safety and Efficacy of Rociletinib in Combination With Trametinib in Patients With mEGFR-positive Advanced or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued development of rociletinib in NSCLC. Stopped enrollment of new patients into all studies involving rociletinib.
Sponsor: Clovis Oncology, Inc. (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-1686-033
Record Dates: First submitted 2015-10-12; First posted 2015-10-20 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — rociletinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rociletinib and Trametinib (Experimental)
  Interventions: Drug: Rociletinib; Drug: Trametinib

INTERVENTIONS:
Drug: Rociletinib
  Other Names: CO-1686
Drug: Trametinib
  Other Names: Mekinist

SUMMARY:
The purpose of this study is to evaluate the safety and anti-tumor effect of rociletinib when administered in combination with trametinib.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, non randomized, multicenter study evaluating the safety and efficacy of rociletinib administered in combination with trametinib.

This study will be conducted in 2 phases:

Phase 1: This will be the dose escalation phase of the study. Phase 1 will determine the MAD or MTD and RP2D of the combination of rociletinib and trametinib, and evaluate its safety and tolerability and PK profile in EGFRm NSCLC patients who have failed at least one prior EGFR TKI.

Phase 2: This will be the dose expansion phase. Phase 2 will evaluate the preliminary efficacy and pharmacodynamics of the combination of rociletinib and trametinib at the RP2D in two subsets of EGFRm NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent on an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved ICF before any study-specific evaluation
* Histologically or cytologically confirmed metastatic or unresectable locally advanced NSCLC with EGFR activating mutation (excluding exon 20 insertion); measurable disease per RECIST 1.1
* Prior treatment with an EGFR TKI; in Phase 2, prior treatment with a T790M-directed EGFR TKI for patients in Group B. Previous chemotherapy is allowed; in Phase 2, immediate prior therapy must be EGFR TKI
* Patient willingness to undergo tumor biopsy at baseline and on treatment (optional for Phase 1; mandatory for Phase 2)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1; life expectancy at least 3 months
* Adequate hematological and biological function; LVEF ≥50%

Exclusion Criteria:

* Documented evidence in tumor of exon 20 insertion, small cell transformation, or MET amplification
* Leptomeningeal carcinomatosis or other untreated or symptomatic CNS metastases (asymptomatic CNS metastases allowed if clinically stable without requirement for steroids within 2 weeks)
* Known preexisting interstitial lung disease or pneumonitis
* Concurrent use of QT-prolonging medication
* Uncontrolled diabetes (HA1C > 10%) despite optional therapy
* Cardiac abnormalities:

  * Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTcF) >450 ms
  * Inability to measure QT interval on ECG
  * Personal or family history of long QT syndrome
  * Implantable pacemaker or implantable cardioverter defibrillator
  * Resting bradycardia < 55 beats/min
* Inability to swallow oral study treatment or any gastrointestinal disease or condition that would preclude adequate absorption of study treatment
* Presence of serious or unstable concomitant systemic disorder incompatible with the clinical study (eg, substance abuse; uncontrolled intercurrent illness including active infection; arterial thrombosis; unstable respiratory, hepatic, renal or cardiac disease; and other active malignancy)
* Pregnant or breastfeeding females and male or female patients who refuse to use adequate contraception during the study and for 16 weeks after the last dose of study treatment
* Any contraindication, allergy, or hypersensitivity to rociletinib, trametinib, or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Continuously, up to approximately 24 months
  Treatment emergent adverse events (AEs), laboratory abnormalities and ECG abnormalities in EGFR-mutant NSCLC patients given oral rociletinib in combination with oral trametinib; defining in Phase 1 the recommended combination dose for further evaluation in Phase 2
Objective Response Rate (ORR) | Every 6 weeks until disease progression, up to approximately 24 months
  ORR according to RECIST Version 1.1 as determined by Investigator assessment
Cmax of rociletinib and trametinib at steady state | Cycle 2 Day 1 to Day 2
Tmax of rociletinib and trametinib at steady state | Cycle 2 Day 1 to Day 2
AUC of rociletinib and trametinib at steady state | Cycle 2 Day 1 to Day 2
Cmin of rociletinib and trametinib at steady state | Cycle 2 Day 1 to Day 2
t1/2 of rociletinib at steady state | Cycle 2 Day 1 to Day 2

SECONDARY OUTCOMES:
Duration of Response (DR) According to RECIST Version 1.1 | Every 6 weeks until disease progression, up to approximately 24 months
  DR according to RECIST Version 1.1 as determined by Investigator assessment
Disease Control Rate (DCR) According to RECIST Version 1.1 | Every 6 weeks until disease progression, up to approximately 24 months
  DCR according to RECIST Version 1.1 as determined by Investigator assessment
Progression Free Survival (PFS) According to RECIST Version 1.1 | Every 6 weeks until disease progression, up to approximately 24 months
  PFS according to RECIST Version 1.1 as determined by Investigator assessment
Overall Survival (OS) | Every 12 weeks until date of death, up to approximately 60 months
Longitudinal changes in blood based biomarkers (i.e. mutations in EGFR) in ctDNA | Biomarker samples will be collected from each subject approximately every 3 weeks, up to approximately 24 months
Cmax of rociletinib metabolites at steady state | Cycle 2 Day 1 to Day 2
Tmax of rociletinib metabolites at steady state | Cycle 2 Day 1 to Day 2
AUC of rociletinib metabolites at steady state | Cycle 2 Day 1 to Day 2
Cmin of rociletinib metabolites at steady state | Cycle 2 Day 1 to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Paula O'Connor, MD, Study Director — Clovis Oncology, Inc.
Locations (4):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
  - Tennessee Oncology, PLLC - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia